CLINICAL TRIAL: NCT02487979
Title: A Phase 2 Study of GPNMB-Targeted Antibody-Drug Conjugate, CDX-011 (Glembatumumab Vedotin, CR011-vcMMAE; NSC# 763737), in Recurrent or Refractory Osteosarcoma
Brief Title: Glembatumumab Vedotin in Treating Patients With Recurrent or Refractory Osteosarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2015-01037; NCI-2015-01037 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AOST1521; s16-01136; AOST1521 (Other: Children's Oncology Group); AOST1521 (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2015-07-01; First posted 2015-07-02 (Estimated); Results first posted 2018-10-15 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Recurrent Osteosarcoma
MeSH Terms: conditions — Osteosarcoma | interventions — glembatumumab vedotin; CR011-vcMMAE

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (glembatumumab vedotin) (Experimental): Patients receive glembatumumab vedotin IV over 90 minutes on day 1. Treatment repeats every 21 days for up to 18 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Glembatumumab Vedotin; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Drug: Glembatumumab Vedotin — Given IV
  Other Names: Antibody-Drug Conjugate CR011-vcMMAE; CDX-011; CR011-vcMMAE; CR011-vcMMAE Immunotoxin
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase II trial studies how well glembatumumab vedotin works in treating patients with osteosarcoma that has come back (recurrent) or does not respond to treatment (refractory). Monoclonal antibodies, such as glembatumumab vedotin, may find tumor cells and help kill them.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate whether CDX-011 (glembatumumab vedotin) therapy either increases the disease control rate at 4 months in patients with recurrent measurable osteosarcoma as compared to an historical Children's Oncology Group (COG) experience or produces an objective response rate in patients without previous eribulin (eribulin mesylate) treatment.

SECONDARY OBJECTIVES:

I. To assess the feasibility and toxicity profile of CDX-011 in patients with recurrent osteosarcoma.

II. To describe the pharmacokinetics of CDX-011 in adolescents and young adults with recurrent osteosarcoma enrolled at COG sites and COG phase I consortium sites only.

III. To determine if there is a relationship between tumor GPNMB expression by immunohistochemistry (IHC) and response to CDX-011 therapy.

IV. To estimate, in the cohort of patients previously treated with eribulin, the proportion who will experience disease progression during the first 4 months of CDX-011 therapy and the proportion of patients who experience a Response Evaluation Criteria in Solid Tumors (RECIST)-defined complete or partial response.

OUTLINE:

Patients receive glembatumumab vedotin intravenously (IV) over 90 minutes on day 1. Treatment repeats every 21 days for up to 18 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have had histologic verification of osteosarcoma at original diagnosis or relapse
* Patients must have measurable disease according to RECIST 1.1, and have relapsed or become refractory to conventional therapy
* Patient must have archival tumor specimen available for submission
* Patients must have a performance status corresponding to Eastern Cooperative Oncology Group (ECOG) scores of 0, 1 or 2; use Karnofsky for patients > 16 years of age and Lansky for patients =< 16 years of age
* Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study

  * Myelosuppressive chemotherapy: must not have received within 2 weeks of entry onto this study (4 weeks if prior nitrosourea)
  * Biologic (anti-neoplastic agent): at least 7 days since the completion of therapy with a biologic agent
  * Radiation therapy (RT): >= 2 weeks for local palliative RT (small port); >= 6 months must have elapsed if prior craniospinal RT or if >= 50% radiation of pelvis; >= 6 weeks must have elapsed if other substantial bone marrow (BM) radiation
  * Monoclonal antibodies: must not have received any monoclonal based therapies within 4 weeks, and all other immunotherapy (tumor vaccine, cytokine, or growth factor given to control the cancer) within 2 weeks, prior to study enrollment
* Peripheral absolute neutrophil count (ANC) >= 1000/uL
* Platelet count >= 75,000/uL (transfusion independent)
* Hemoglobin >= 8.0 g/dL (may receive red blood cell [RBC] transfusions)
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2 or a serum creatinine based on age/gender as follows:

  * Age 1 to < 2 years (male and female: 0.6 mg/dL)
  * Age 2 to < 6 years (male and female: 0.8 mg/dL)
  * Age 6 to < 10 years (male and female: 1 mg/dL)
  * Age 10 to < 13 years (male and female: 1.2 mg/dL)
  * Age 13 to < 16 years (male: 1.5 mg/dL and female: 1.4 mg/dL)
  * Age >= 16 (male: 1.7 mg/dL and female: 1.4 mg/dL)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) for age
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) or serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) < 110 U/L; for the purposes of this study the ULN for SGPT is defined as 45 U/L
* Serum albumin > 2 g/dL
* Shortening fraction of >= 27% by echocardiogram, or
* Ejection fraction of >= 50% by radionuclide angiogram
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Exclusion Criteria:

* Patients with > grade 2 neuropathy according to the Modified ("Balis") Pediatric Scale of Peripheral Neuropathies will be excluded except in cases in which neuropathy is secondary to prior surgery
* Patients who have previously received CDX-011 (CR011-vc monomethyl auristatin E [MMAE]; CDX-011) or other MMAE-containing agents
* Patients who have received other investigational drugs within 2 weeks or 5 half-lives (whichever is longer) prior to study enrollment
* Patients with a history of allergic reactions attributed to compounds of similar composition to dolastatin or auristatin; compounds of similar composition include auristatin PHE as an anti-fungal agent, auristatin PE (TZT-1027, Soblidotin, NSC-654663) as an anti-tumor agent and symplostatin 1 as an anti-tumor agent
* Patients with known central nervous system metastasis are not eligible
* Patients who have had major surgery within 2 weeks prior to enrollment are not eligible; procedures such as placement of a central vascular catheter, or limited tumor biopsy, are not considered major surgery
* Female patients who are pregnant are ineligible
* Lactating females are not eligible unless they have agreed not to breastfeed their infants
* Female patients of childbearing potential are not eligible unless a negative pregnancy test result has been obtained
* Sexually active patients of reproductive potential are not eligible unless they have agreed to use an effective contraceptive method for the duration of their study participation and for 2 months after the end of study treatment

Ages: 12 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2016-02-16 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M Kopp, Principal Investigator — Children's Oncology Group
Locations (155):
- United States (149):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - PCR Oncology, Arroyo Grande, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Kaiser Permanente-Capitol Hill Medical Center, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Hospital, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - IU Health North Hospital, Carmel, Indiana
  - Riley Hospital for Children, Indianapolis, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - 21st Century Oncology-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - 21st Century Oncology, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - 21st Century Oncology-Vegas Tenaya, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - 21st Century Oncology-Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Albany Medical Center, Albany, New York
  - NYU Winthrop Hospital, Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Children's Hospital at Montefiore, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Oncology Group, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Vanderbilt-Ingram Cancer Center Cool Springs, Franklin, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Cancer Therapy and Research Center at The UT Health Science Center at San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University Hospital, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Canada (5):
  - Alberta Children's Hospital, Calgary, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec
- University Pediatric Hospital, San Juan, Puerto Rico

REFERENCES:
- [Derived] Kopp LM, Malempati S, Krailo M, Gao Y, Buxton A, Weigel BJ, Hawthorne T, Crowley E, Moscow JA, Reid JM, Villalobos V, Randall RL, Gorlick R, Janeway KA. Phase II trial of the glycoprotein non-metastatic B-targeted antibody-drug conjugate, glembatumumab vedotin (CDX-011), in recurrent osteosarcoma AOST1521: A report from the Children's Oncology Group. Eur J Cancer. 2019 Nov;121:177-183. doi: 10.1016/j.ejca.2019.08.015. Epub 2019 Oct 3. PMID 31586757
- [Derived] Hattinger CM, Patrizio MP, Magagnoli F, Luppi S, Serra M. An update on emerging drugs in osteosarcoma: towards tailored therapies? Expert Opin Emerg Drugs. 2019 Sep;24(3):153-171. doi: 10.1080/14728214.2019.1654455. Epub 2019 Aug 14. PMID 31401903

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Glembatumumab Vedotin)
Started | 22
Completed | 1
Not Completed | 21
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 2
Not completed — Progressive Disease | 17

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Glembatumumab Vedotin)
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.09 (5.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Canada | 1
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Disease Control Success
Description: The number of patients who do not experience disease progression or death in the six cycles following enrollment on AOST1521
Time Frame: First six cycles (21-day cycle) of protocol therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Glembatumumab Vedotin)
Number analyzed (Participants) | 22
Participants | 3

2. Secondary Outcome: Toxicity Associated With Chemotherapy
Description: The number of cycles aggregated across all patients where CTC Version 4 grade 3 or higher.
Time Frame: Duration of protocol therapy - Up to two years
Population: 22 patients were treated on protocol therapy. Sixty-one (61) cycles were reported for the analysis of toxicity.
Measure: Number; unit: cycles
Arm/Group | Treatment (Glembatumumab Vedotin)
Number analyzed (Participants) | 22
cycles
  Incidence of Abdominal Pain | 2
  Incidence of acneiform rash | 1
  Incidence of Anaphylaxis | 1
  Incidence of Anemia | 2
  Incidence of Anorexia | 1
  Incidence of Back Pain | 2
  Incidence of Constipation | 1
  Incidence of Febrile Neutropenia | 1
  Incidence of Headache | 1
  Incidence of Hypertension | 1
  Incidence of Hypocalcemia | 1
  Incidence of Hypokalemia | 4
  Incidence of Hypophosphatemia | 2
  Incidence of Hypotension | 1
  Incidence of Leukopenia | 1
  Incidence of Lymphopenia | 1
  Incidence of Mucocitis | 2
  Incidence of Myalgia | 1
  Incidence of Nausea | 1
  Incidence of Neutropenia | 2
  Incidence of Pain | 2
  Incidence of Pneumothorax | 1
  Incidence of Thrombocytopenia | 1

3. Secondary Outcome: Pharmacokinetics of Glembatumumab Vedotin: Total Antibody and Antibody-drug Conjugate Half-life
Description: Total antibody and antibody-drug conjugate half-life are estimated from the sampling time points: Before first dose (Baseline), end of infusion, at 1, 2, 4, and 24 hours post infusion
Time Frame: Baseline to 24 hours post infusion on course 1
Population: Samples were provided for four patients
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Treatment (Glembatumumab Vedotin)
Number analyzed (Participants) | 4
hours
  Total antibody half-life | 35.2 (6.4)
  Antibody-Drug Conjugate half-life | 29.1 (8.4)

4. Secondary Outcome: Pharmacokinetics of Glembatumumab Vedotin: Total Antibody and Antibody-drug Conjugate Clearance
Description: Total antibody and antibody-drug conjugate clearance are estimated from the sampling time points: Before first dose (Baseline), end of infusion, at 1, 2, 4, and 24 hours post infusion
Time Frame: Baseline to 24 hours post infusion on course 1
Population: Samples were provided for four patients
Measure: Mean (Standard Deviation); unit: millilitres per hour per kilogram
Arm/Group | Treatment (Glembatumumab Vedotin)
Number analyzed (Participants) | 4
millilitres per hour per kilogram
  Total antibody clearance | 0.8 (0.1)
  Antibody-Drug Conjugate clearance | 0.9 (0.3)

5. Secondary Outcome: Pharmacokinetics of Glembatumumab Vedotin: Total Antibody and Antibody-drug Conjugate Areas Under the Curve
Description: Total antibody and antibody-drug conjugate areas under the curve are estimated from the sampling time points: Before first dose (Baseline), end of infusion, at 1, 2, 4, and 24 hours post infusion
Time Frame: Baseline to 24 hours post infusion on course 1
Population: Samples were provided for four patients
Measure: Mean (Standard Deviation); unit: hour-microgram per millilitre
Arm/Group | Treatment (Glembatumumab Vedotin)
Number analyzed (Participants) | 4
hour-microgram per millilitre
  Total antibody area under the curve | 2320.0 (342)
  Antibody-Drug Conjugate area under the curve | 2259.5 (749.6)

6. Secondary Outcome: Number of Participants With Glycoprotein NMB (GPNMB) Expression Stratified by Immunohistochemistry (IHC) Staining Strength
Description: GPNMB expression by IHC of 0+ to 3+ staining strength as assessed on archived tumor specimens. 0 being no GPNMB expression and 3 indicating strong GPNMB expression.
Time Frame: Prior to the time of enrollment
Population: Analysis was successfully completed for 19 patients
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Glembatumumab Vedotin)
Number analyzed (Participants) | 19
Participants
  0+ staining strength | 1
  1+ staining strength | 3
  2+ staining strength | 2
  3+ staining strength | 13

7. Secondary Outcome: RECIST Response
Description: The number of patients who experience a complete or partial response according the RECIST criteria for target lesions complete response (CR) disappearance of all lesions; partial response (PR ) >= 30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR+PR.
Time Frame: First six cycles (21-day cycle) of protocol therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Glembatumumab Vedotin)
Number analyzed (Participants) | 22
Participants | 1

ADVERSE EVENTS:
Time Frame: Overall protocol therapy up to 14 months in total or 18 cycles, whichever occurs first.
Description: Adverse event reporting is collected routinely using case report forms. SAE field contains NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted via expedited reporting (NCI AdEERs / CAeRs). The AE field contains grade 3 and higher CTCAEs reported on study excluding those that were reported as SAEs. Ineligible patients are excluded from reporting of adverse events.
Arm/Group | Treatment (Glembatumumab Vedotin)
All-Cause Mortality (participants affected / at risk) | 14/22
Serious Adverse Events (participants affected / at risk) | 8/22
Other Adverse Events (participants affected / at risk) | 7/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Glembatumumab Vedotin) (N=22)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Anaphylaxis (Immune system disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Glembatumumab Vedotin) (N=22)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
Hypertension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-06): https://cdn.clinicaltrials.gov/large-docs/79/NCT02487979/Prot_SAP_000.pdf